CLINICAL TRIAL: NCT03462173
Title: A Phase I, Randomized，Double-blind, Placebo-controlled, Single Ascending Dose, Single-center Study to Assess the Safety, Tolerability and Pharmacokinetic of Yimitasvir in Healthy Adults Subjects
Brief Title: The Safety, Tolerability and Pharmacokinetic Study of Yimitasvir in Healthy Adults Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCD-DDAG181PA-13-001
Record Dates: First submitted 2018-02-09; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — yimitasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 30 mg single dose (Experimental): Healthy subjects, receiving a single dose of 30 mg yimitasvir(N=6) or placebo(N=2)
  Interventions: Drug: yimitasvir; Drug: placebo
- 100 mg single dose (Experimental): Healthy subjects, receiving a single dose of 100 mg yimitasvir (N=6) or placebo(N=2)
  Interventions: Drug: yimitasvir; Drug: placebo
- 200 mg single dose (Experimental): Healthy subjects, receiving a single dose of 200 mg yimitasvir (N=6) or placebo(N=2)
  Interventions: Drug: yimitasvir; Drug: placebo
- 400 mg single dose (Experimental): Healthy subjects, receiving a single dose of 400 mg yimitasvir (N=6) or placebo(N=2)
  Interventions: Drug: yimitasvir; Drug: placebo
- 600 mg single dose (Experimental): Healthy subjects, receiving a single dose of 600 mg yimitasvir (N=6) or placebo(N=2)
  Interventions: Drug: yimitasvir; Drug: placebo
- 800 mg single dose (Experimental): Healthy subjects, receiving a single dose of 800 mg yimitasvir (N=6) or placebo(N=2)
  Interventions: Drug: yimitasvir; Drug: placebo
- 1000 mg single dose (Experimental): Healthy subjects, receiving a single dose of 1000 mg yimitasvir (N=6) or placebo(N=2)
  Interventions: Drug: yimitasvir; Drug: placebo

INTERVENTIONS:
Drug: yimitasvir — Capsule administered orally once daily
  Other Names: DAG181
Drug: placebo — Matching Placebo Capsule
  Other Names: DAG181 placebo

SUMMARY:
The Safety, Tolerability and Pharmacokinetic Study of Chronic Hepatitis C Treatment Drug Yimitasvir in Healthy Adults Subjects.

DETAILED DESCRIPTION:
This was a Randomized，Double-blind, Placebo-controlled, Single Ascending Dose, Single-center Study to Assess the Safety, Tolerability and Pharmacokinetic of Yimitasvir in Healthy Adults Subjects

A total of 56 healthy subjects were divided into 7 groups, with each group consisting of 8 subjects. Six of the subjects received the investigational drug, and two received placebo. All of the subjects received a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, overall healthy subjects;
* Between 18 and 45 years of age, inclusive, similar ages;
* Body weight should be≥50 kg; Body Mass Index (BMI) is between 19 and 25 kg/m2, inclusive, similar body weights;
* Able to comprehend and sign the ICF voluntarily prior to initiate the study;
* Able to communicate well with the investigator and complete the study according to the protocol.

Exclusion Criteria:

* Pregnant or nursing female, or plan for pregnancy within 6 months;
* Female with positive urine pregnancy test results;
* Positive test results for HBsAg, anti-HCV Ab, anti-HIV Ab or syphilis;
* Have taken any drug inhibiting gastric acid secretion within 1 month prior to study drug administration, such as: H2 receptor antagonists (eg: Cimetidine, Ranitidine, Famotidine, Nizatidine and Roxatidine); Proton pump inhibitors (eg: Omeprazole, Lansoprazole, Rabeprazole, Pantoprazole and Esomeprazole); cholinoceptor blocking drugs (eg: Atropine and Pirenzepine);
* History of immune system disease (such as thymus disease);
* Have undergone major surgery within 6 months before enrollment;
* History of tumor;
* Drink frequently within 6 months prior to study drug administration, namely alcohol consumption are more than 20 grams per day;
* Smokers, who smoke more than 1 cigarettes/day within 3 months before the study;
* Participated in any clinical trial within 3 months prior to the study;
* Cannot be tolerant to oral drugs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2016-01-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | Baseline to day 10
  To assess the safety and tolerability after a single dose of DAG181
Cmax | Prior to dosing (0 h) and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 h after dosing
  Maximum observed plasma concentration of DAG181
Tmax | Prior to dosing (0 h) and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 h after dosing
  Time of the maximum observed plasma concentration
AUC | Prior to dosing (0 h) and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 h after dosing
  Area under the plasma concentration-time curve (AUC)
T1/2 | Prior to dosing (0 h) and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 h after dosing
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Cui, Doctor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No